CLINICAL TRIAL: NCT00345839
Title: EValuation Of Cinacalcet Hydrochloride (HCl) Therapy to Lower CardioVascular Events
Brief Title: E.V.O.L.V.E. Trial™: EValuation Of Cinacalcet Hydrochloride (HCl) Therapy to Lower CardioVascular Events
Acronym: EVOLVE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20050182
Record Dates: First submitted 2006-06-27; First posted 2006-06-29 (Estimated); Results first posted 2014-01-22 (Estimated); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Secondary Hyperparathyroidism; Chronic Kidney Disease
Keywords: Cinacalcet HCl; Cinacalcet; AMG 073; Sensipar; Mimpara; Calcimimetic; Hemodialysis; CKD; Secondary hyperparathyroidism (HPT)
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Renal Insufficiency, Chronic | interventions — Cinacalcet

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cinacalcet (Experimental)
  Interventions: Drug: Cinacalcet
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cinacalcet — Possible doses: 30, 60, 90, 120, and 180 mg using tablet strengths of 30, 60, or 90 mg. Sequential titration starting at 30 mg daily (QD), once every 4 weeks for the first 20 weeks and once every 8 weeks after Week 20. Titration increases or decreases based on PTH values, serum calcium, and safety. Daily dosing unless temporary hold criteria or withdrawal criteria is met, or until study completion; estimated 2.5 to 4 years of intervention.
  Arms: Cinacalcet
Drug: Placebo — Possible doses: 30, 60, 90, 120, and 180 mg using tablet strengths of 30, 60, or 90 mg. Sequential titration starting at 30 mg QD, once every 4 weeks for the first 20 weeks and once every 8 weeks after Week 20. Titration increases or decreases based on PTH values, serum calcium, and safety. Daily dosing unless temporary hold criteria or withdrawal criteria is met, or until study completion; estimated 2.5 to 4 years of intervention.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effects of cinacalcet (cinacalcet HCl or Sensipar®/Mimpara®) on cardiovascular events and death in chronic kidney disease (CKD) patients with secondary hyperparathyroidism (HPT) who are receiving dialysis.

DETAILED DESCRIPTION:
Secondary HPT is common in people with CKD. Patients with secondary HPT often have high parathyroid hormone (PTH) levels and may develop large parathyroid glands in the neck. Patients with secondary HPT may have bone disease (osteodystrophy). This bone disease may cause bone pain, fractures, and poor formation of red blood cells. Other problems from secondary HPT may include increases in blood levels of calcium and phosphorus. These may cause calcium to deposit in body tissues. Calcium deposits can cause arthritis (joint pain and swelling), muscle inflammation, itching, gangrene (death of soft tissue), or heart and lung problems. New evidence suggests that secondary HPT is associated with cardiovascular disease and increased death risk. The purpose of this study is to evaluate the effects of cinacalcet (cinacalcet HCl or Sensipar®/Mimpara®) on cardiovascular events (having to do with the heart and its blood vessels) and death in chronic kidney disease (CKD) patients with secondary hyperparathyroidism (HPT) who are receiving dialysis. These events include death from any reason, heart attack and episodes where the heart does not get enough oxygen, peripheral vascular disease (narrowing of vessels that carry blood to the legs, arms, stomach or kidneys), and heart failure (a condition that occurs when the heart is unable to pump enough blood to meet the need's of the body's tissues)

ELIGIBILITY:
Inclusion Criteria:

* Inclusion:≥ 18 years of age
* Treated with maintenance hemodialysis - PTH ≥ 300 pg/mL (31.8 pmol/L)
* serum calcium ≥ 8.4mg/dL (2.1 mmol/L)
* Ca x P ≥ 45 mg2*/dL2 (3.63 mmol2/L2)

Exclusion Criteria: - Exclusion:

* Parathyroidectomy in the 12 weeks before the date of informed consent
* Received therapy with cinacalcet within 3 months of randomization
* Hospitalization within 12 weeks of randomization for any of the following events: a. Myocardial ischemia b. Unstable angina c. Heart Failure (HF) (including any unplanned presentation to a health care facility that would require mechanical intervention [i.e., unplanned dialysis treatment]) d. Peripheral vascular disease (other than dialysis vascular access revision) e. Stroke
* History of seizure within 12 weeks prior to randomization
* Scheduled date for kidney transplant from a known living donor
* Anticipated parathyroidectomy within 6 months after randomization

  * in all instances, the 2 refers to squared.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3883 (Actual)
Dates: Start 2006-08-22 (Actual); Primary Completion 2012-04-10 (Actual); Study Completion 2012-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Chertow GM, Correa-Rotter R, Block GA, Drueke TB, Floege J, Goodman WG, Herzog CA, Kubo Y, London GM, Mahaffey KW, Mix TC, Moe SM, Wheeler DC, Parfrey PS. Baseline characteristics of subjects enrolled in the Evaluation of Cinacalcet HCl Therapy to Lower Cardiovascular Events (EVOLVE) trial. Nephrol Dial Transplant. 2012 Jul;27(7):2872-9. doi: 10.1093/ndt/gfr777. Epub 2012 Apr 23. PMID 22529163
- [Background] Chertow GM, Pupim LB, Block GA, Correa-Rotter R, Drueke TB, Floege J, Goodman WG, London GM, Mahaffey KW, Moe SM, Wheeler DC, Albizem M, Olson K, Klassen P, Parfrey P. Evaluation of Cinacalcet Therapy to Lower Cardiovascular Events (EVOLVE): rationale and design overview. Clin J Am Soc Nephrol. 2007 Sep;2(5):898-905. doi: 10.2215/CJN.04381206. Epub 2007 Aug 16. PMID 17702710
- [Background] EVOLVE Trial Investigators; Chertow GM, Block GA, Correa-Rotter R, Drueke TB, Floege J, Goodman WG, Herzog CA, Kubo Y, London GM, Mahaffey KW, Mix TC, Moe SM, Trotman ML, Wheeler DC, Parfrey PS. Effect of cinacalcet on cardiovascular disease in patients undergoing dialysis. N Engl J Med. 2012 Dec 27;367(26):2482-94. doi: 10.1056/NEJMoa1205624. Epub 2012 Nov 3. PMID 23121374
- [Background] Parfrey PS, Chertow GM, Block GA, Correa-Rotter R, Drueke TB, Floege J, Herzog CA, London GM, Mahaffey KW, Moe SM, Wheeler DC, Dehmel B, Trotman ML, Modafferi DM, Goodman WG. The clinical course of treated hyperparathyroidism among patients receiving hemodialysis and the effect of cinacalcet: the EVOLVE trial. J Clin Endocrinol Metab. 2013 Dec;98(12):4834-44. doi: 10.1210/jc.2013-2975. Epub 2013 Oct 9. PMID 24108314
- [Derived] Floege J, Tsirtsonis K, Iles J, Drueke TB, Chertow GM, Parfrey P. Incidence, predictors and therapeutic consequences of hypocalcemia in patients treated with cinacalcet in the EVOLVE trial. Kidney Int. 2018 Jun;93(6):1475-1482. doi: 10.1016/j.kint.2017.12.014. Epub 2018 Mar 7. PMID 29525393
- [Derived] Abdalla S, Montez-Rath ME, Parfrey PS, Chertow GM. The win ratio approach to analyzing composite outcomes: An application to the EVOLVE trial. Contemp Clin Trials. 2016 May;48:119-24. doi: 10.1016/j.cct.2016.04.001. Epub 2016 Apr 11. PMID 27080930
- [Derived] Moe SM, Chertow GM, Parfrey PS, Kubo Y, Block GA, Correa-Rotter R, Drueke TB, Herzog CA, London GM, Mahaffey KW, Wheeler DC, Stolina M, Dehmel B, Goodman WG, Floege J; Evaluation of Cinacalcet HCl Therapy to Lower Cardiovascular Events (EVOLVE) Trial Investigators*. Cinacalcet, Fibroblast Growth Factor-23, and Cardiovascular Disease in Hemodialysis: The Evaluation of Cinacalcet HCl Therapy to Lower Cardiovascular Events (EVOLVE) Trial. Circulation. 2015 Jul 7;132(1):27-39. doi: 10.1161/CIRCULATIONAHA.114.013876. Epub 2015 Jun 9. PMID 26059012
- [Derived] Floege J, Kubo Y, Floege A, Chertow GM, Parfrey PS. The Effect of Cinacalcet on Calcific Uremic Arteriolopathy Events in Patients Receiving Hemodialysis: The EVOLVE Trial. Clin J Am Soc Nephrol. 2015 May 7;10(5):800-7. doi: 10.2215/CJN.10221014. Epub 2015 Apr 17. PMID 25887067
- [Derived] Kubo Y, Sterling LR, Parfrey PS, Gill K, Mahaffey KW, Gioni I, Trotman ML, Dehmel B, Chertow GM. Assessing the treatment effect in a randomized controlled trial with extensive non-adherence: the EVOLVE trial. Pharm Stat. 2015 May-Jun;14(3):242-51. doi: 10.1002/pst.1680. Epub 2015 Apr 6. PMID 25851955
- [Derived] Parfrey PS, Drueke TB, Block GA, Correa-Rotter R, Floege J, Herzog CA, London GM, Mahaffey KW, Moe SM, Wheeler DC, Kubo Y, Dehmel B, Goodman WG, Chertow GM; Evaluation of Cinacalcet HCl Therapy to Lower Cardiovascular Events (EVOLVE) Trial Investigators. The Effects of Cinacalcet in Older and Younger Patients on Hemodialysis: The Evaluation of Cinacalcet HCl Therapy to Lower Cardiovascular Events (EVOLVE) Trial. Clin J Am Soc Nephrol. 2015 May 7;10(5):791-9. doi: 10.2215/CJN.07730814. Epub 2015 Feb 20. PMID 25710802
- [Derived] Wheeler DC, London GM, Parfrey PS, Block GA, Correa-Rotter R, Dehmel B, Drueke TB, Floege J, Kubo Y, Mahaffey KW, Goodman WG, Moe SM, Trotman ML, Abdalla S, Chertow GM, Herzog CA; EValuation Of Cinacalcet HCl Therapy to Lower CardioVascular Events (EVOLVE) Trial Investigators. Effects of cinacalcet on atherosclerotic and nonatherosclerotic cardiovascular events in patients receiving hemodialysis: the EValuation Of Cinacalcet HCl Therapy to Lower CardioVascular Events (EVOLVE) trial. J Am Heart Assoc. 2014 Nov 17;3(6):e001363. doi: 10.1161/JAHA.114.001363. PMID 25404192
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from dialysis clinics and hospitals between August 2006 to Jan 2008 from 22 countries.
Pre-assignment Details: Participants were screened over a 30 day period.
Groups:
- Cinacalcet: Cinacalcet administered orally in doses of 30, 60, 90, 120 or 180 mg per day. Participants could be titrated up to maximum dose based on PTH (parathyroid hormone), serum calcium and safety assessments.
- Placebo: Participants were given matching placebo tablets compared to the cinacalcet group.
Period: Overall Study
Arm/Group | Cinacalcet | Placebo
Started | 1948 (Randomized to cinacalcet) | 1935 (Randomized to placebo)
Completed | 1799 (Participants who completed study includes those with ended study due to death.) | 1776 (Participants who completed study includes those with ended study due to death.)
Not Completed | 149 | 159
Not completed — Withdrawal by Subject | 91 | 98
Not completed — Lost to Follow-up | 58 | 61

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cinacalcet | Placebo | Total
Number analyzed (Participants) | 1948 | 1935 | 3883
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.8 (14.5) | 54.0 (14.2) | 54.4 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 809 | 769 | 1578
  Male | 1139 | 1166 | 2305
Race/Ethnicity, Customized [Number; unit: Participants]
  White or Caucasian | 1124 | 1116 | 2240
  Black or African American | 409 | 428 | 837
  Hispanic or Latino | 317 | 310 | 627
  Asian | 47 | 38 | 85
  Japanese | 4 | 1 | 5
  American Indian or Alaska Native | 5 | 7 | 12
  Native Hawaiian or Other Pacific Islander | 12 | 9 | 21
  Aborigine | 1 | 4 | 5
  Other | 29 | 22 | 51
History of Diabetes Stratification Factor [Number; unit: Participants] — History of diabetes stratification factor from the interactive voice response system.
  Participants
    Diabetes | 619 | 614 | 1233
    No Diabetes | 1329 | 1321 | 2650
Country stratification factor [Number; unit: Participants] — Country stratification factor from the interactive voice response system. Denmark and Sweden were combined to create Nordic stratum.
  Participants
    Argentina | 171 | 170 | 341
    Australia | 74 | 75 | 149
    Austria | 31 | 29 | 60
    Belgium | 50 | 50 | 100
    Brazil | 151 | 150 | 301
    Canada | 73 | 73 | 146
    Denmark | 8 | 11 | 19
    France | 40 | 40 | 80
    Germany | 81 | 81 | 162
    Hungary | 66 | 67 | 133
    Ireland | 5 | 6 | 11
    Italy | 69 | 68 | 137
    Mexico | 23 | 22 | 45
    Netherlands | 15 | 14 | 29
    Poland | 59 | 57 | 116
    Portugal | 22 | 21 | 43
    Russia | 143 | 140 | 283
    Spain | 40 | 38 | 78
    Sweden | 13 | 10 | 23
    Switzerland | 18 | 19 | 37
    United Kingdom | 81 | 79 | 160
    United States | 715 | 715 | 1430

OUTCOME MEASURES:

1. Primary Outcome: Time to Primary Composite Endpoint (All-cause Mortality, Myocardial Infarction, Hospitalization for Unstable Angina, Heart Failure or Peripheral Vascular Event)
Description: Time to Primary Composite Endpoint (All-cause Mortality, Myocardial Infarction, Hospitalization for Unstable Angina, Heart Failure or Peripheral Vascular Event). Stratified by history of diabetes and country.
Time Frame: From date of randomization until date of first confirmed primary composite endpoint event, assessed up to 5.4 years
Population: Utilizes the Efficacy Analysis Set which includes all randomized participants. Participants were analyzed in the treatment group as randomized using the Intent-to-treat (ITT) method.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Cinacalcet | Placebo
Number analyzed (Participants) | 1948 | 1935
Months | 55.0 [22.6 to NA] — NA (Not Applicable) indicates that the parameter is not estimable due to insufficient number of subjects with events. | 53.0 [19.1 to NA] — NA (Not Applicable) indicates that the parameter is not estimable due to insufficient number of subjects with events.
Statistical Analysis 1: Comparison: Cinacalcet vs Placebo; Test type: Superiority or Other; p = 0.112, Log Rank — p-value<0.044 considered significant; Stratified by history of diabetes and country. 2-sided test
Statistical Analysis 2: Comparison: Cinacalcet vs Placebo; Test type: Superiority or Other; Regression, Cox; Stratified by history of diabetes and country; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.85 to 1.02] — HR is cinacalcet vs placebo

2. Secondary Outcome: Time to All-cause Mortality
Description: Time to All-cause Mortality. Stratified by history of diabetes and country.
Time Frame: From date of randomization until date of confirmed all-cause mortality endpoint event, assessed up to 5.4 years
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Cinacalcet | Placebo
Number analyzed (Participants) | 1948 | 1935
Months | NA [37.9 to NA] — NA (Not Applicable) indicates that the parameter is not estimable due to insufficient number of subjects with events. | NA [31.6 to NA] — NA (Not Applicable) indicates that the parameter is not estimable due to insufficient number of subjects with events.
Statistical Analysis 1: Comparison: Cinacalcet vs Placebo; Test type: Superiority or Other; p = 0.249, Log Rank — No adjustments for multiple comparisons were made for the components of the primary composite endpoint since the purpose of these analyses is to show how each component contributes to the results of the composite; Stratified by history of diabetes and country. 2-sided test
Statistical Analysis 2: Comparison: Cinacalcet vs Placebo; Test type: Superiority or Other; Regression, Cox; Stratified by history of diabetes and country; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.85 to 1.04] — HR is cinacalcet vs placebo

3. Secondary Outcome: Time to Myocardial Infarction
Description: Time to Myocardial Infarction. Stratified by history of diabetes and country.
Time Frame: From date of randomization until date of first confirmed myocardial infarction endpoint event, assessed up to 5.4 years
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Cinacalcet | Placebo
Number analyzed (Participants) | 1948 | 1935
Months | NA [NA to NA] — NA (Not Applicable) indicates that the parameter is not estimable due to insufficient number of subjects with events. | NA [NA to NA] — NA (Not Applicable) indicates that the parameter is not estimable due to insufficient number of subjects with events.
Statistical Analysis 1: Comparison: Cinacalcet vs Placebo; Test type: Superiority or Other; p = 0.800, Log Rank — [p-value comment as in outcome 2, analysis 1]; Stratified by history of diabetes and country. 2-sided test
Statistical Analysis 2: Comparison: Cinacalcet vs Placebo; Test type: Superiority or Other; Regression, Cox; Stratified by history of diabetes and country; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.79 to 1.19] — HR is cinacalcet vs placebo

4. Secondary Outcome: Time to Hospitalization for Unstable Angina
Description: Time to Hospitalization for Unstable Angina. Stratified by history of diabetes and country.
Time Frame: From date of randomization until date of first confirmed hospitalization for unstable angina endpoint event, assessed up to 5.4 years
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Cinacalcet | Placebo
Number analyzed (Participants) | 1948 | 1935
Months | NA [NA to NA] — NA (Not Applicable) indicates that the parameter is not estimable due to insufficient number of subjects with events. | NA [NA to NA] — NA (Not Applicable) indicates that the parameter is not estimable due to insufficient number of subjects with events.
Statistical Analysis 1: Comparison: Cinacalcet vs Placebo; Test type: Superiority or Other; p = 0.283, Log Rank — [p-value comment as in outcome 2, analysis 1]; Stratified by history of diabetes and country. 2-sided test
Statistical Analysis 2: Comparison: Cinacalcet vs Placebo; Test type: Superiority or Other; Regression, Cox; Stratified by history of diabetes and country; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.58 to 1.18] — HR is cinacalcet vs placebo

5. Secondary Outcome: Time to Heart Failure
Description: Time to Heart Failure. Stratified by history of diabetes and country.
Time Frame: From date of randomization until date of first confirmed heart failure endpoint event, assessed up to 5.4 years
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Cinacalcet | Placebo
Number analyzed (Participants) | 1948 | 1935
Months | NA [NA to NA] — NA (Not Applicable) indicates that the parameter is not estimable due to insufficient number of subjects with events. | NA [NA to NA] — NA (Not Applicable) indicates that the parameter is not estimable due to insufficient number of subjects with events.
Statistical Analysis 1: Comparison: Cinacalcet vs Placebo; Test type: Superiority or Other; p = 0.034, Log Rank — [p-value comment as in outcome 2, analysis 1]; Stratified by history of diabetes and country. 2-sided test
Statistical Analysis 2: Comparison: Cinacalcet vs Placebo; Test type: Superiority or Other; Regression, Cox; Stratified by history of diabetes and country; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.68 to 0.99] — HR is cinacalcet vs placebo

6. Secondary Outcome: Time to Peripheral Vascular Event
Description: Time to Peripheral Vascular Event. Stratified by history of diabetes and country.
Time Frame: From date of randomization until date of first confirmed peripheral vascular endpoint event, assessed up to 5.4 years
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Cinacalcet | Placebo
Number analyzed (Participants) | 1948 | 1935
Months | NA [NA to NA] — NA (Not Applicable) indicates that the parameter is not estimable due to insufficient number of subjects with events. | NA [NA to NA] — NA (Not Applicable) indicates that the parameter is not estimable due to insufficient number of subjects with events.
Statistical Analysis 1: Comparison: Cinacalcet vs Placebo; Test type: Superiority or Other; p = 0.190, Log Rank — [p-value comment as in outcome 2, analysis 1]; Stratified by history of diabetes and country. 2-sided test
Statistical Analysis 2: Comparison: Cinacalcet vs Placebo; Test type: Superiority or Other; Regression, Cox; Stratified by history of diabetes and country; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.72 to 1.07] — HR is cinacalcet vs placebo

7. Secondary Outcome: Time to Cardiovascular Mortality
Description: Time to Cardiovascular Mortality. Stratified by history of diabetes and country.
Time Frame: From date of randomization until date of first confirmed cardiovascular mortality endpoint event, assessed up to 5.4 years
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Cinacalcet | Placebo
Number analyzed (Participants) | 1948 | 1935
Months | NA [NA to NA] — NA (Not Applicable) indicates that the parameter is not estimable due to insufficient number of subjects with events. | NA [NA to NA] — NA (Not Applicable) indicates that the parameter is not estimable due to insufficient number of subjects with events.
Statistical Analysis 1: Comparison: Cinacalcet vs Placebo; Test type: Superiority or Other; p = 0.277, Log Rank — No adjustments for multiple comparisons were made for this endpoint; Stratified by history of diabetes and country. 2-sided test
Statistical Analysis 2: Comparison: Cinacalcet vs Placebo; Test type: Superiority or Other; Regression, Cox; Stratified by history of diabetes and country; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.80 to 1.07] — HR is cinacalcet vs placebo

8. Secondary Outcome: Time to Stroke
Description: Time to Stroke. Stratified by history of diabetes and country.
Time Frame: From date of randomization until date of first confirmed stroke endpoint event, assessed up to 5.4 years
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Cinacalcet | Placebo
Number analyzed (Participants) | 1948 | 1935
Months | NA [NA to NA] — NA (Not Applicable) indicates that the parameter is not estimable due to insufficient number of subjects with events. | NA [NA to NA] — NA (Not Applicable) indicates that the parameter is not estimable due to insufficient number of subjects with events.
Statistical Analysis 1: Comparison: Cinacalcet vs Placebo; Test type: Superiority or Other; p = 0.607, Log Rank — No adjustments for multiple comparisons were made for this endpoint; Stratified by history of diabetes and country. 2-sided test
Statistical Analysis 2: Comparison: Cinacalcet vs Placebo; Test type: Superiority or Other; Regression, Cox; Stratified by history of diabetes and country; Hazard Ratio (HR) = 1.07, 95% CI 2-sided [0.82 to 1.40] — HR is cinacalcet vs placebo

9. Secondary Outcome: Time to Bone Fracture
Description: Time to Bone Fracture. Stratified by history of diabetes and country.
Time Frame: From date of randomization until date of first confirmed bone fracture endpoint event, assessed up to 5.4 years
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Cinacalcet | Placebo
Number analyzed (Participants) | 1948 | 1935
Months | NA [NA to NA] — NA (Not Applicable) indicates that the parameter is not estimable due to insufficient number of subjects with events. | NA [NA to NA] — NA (Not Applicable) indicates that the parameter is not estimable due to insufficient number of subjects with events.
Statistical Analysis 1: Comparison: Cinacalcet vs Placebo; Test type: Superiority or Other; p = 0.218, Log Rank — No adjustments for multiple comparisons were made for this endpoint; Stratified by history of diabetes and country. 2-sided test
Statistical Analysis 2: Comparison: Cinacalcet vs Placebo; Test type: Superiority or Other; Regression, Cox; Stratified by history of diabetes and country; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.75 to 1.07] — HR is cinacalcet vs placebo

10. Secondary Outcome: Time to Parathyroidectomy
Description: Time to Parathyroidectomy. Stratified by history of diabetes and country.
Time Frame: From date of randomization until date of first confirmed parathyroidectomy endpoint event, assessed up to 5.4 years
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Cinacalcet | Placebo
Number analyzed (Participants) | 1948 | 1935
Months | NA [NA to NA] — NA (Not Applicable) indicates that the parameter is not estimable due to insufficient number of subjects with events. | NA [NA to NA] — NA (Not Applicable) indicates that the parameter is not estimable due to insufficient number of subjects with events.
Statistical Analysis 1: Comparison: Cinacalcet vs Placebo; Test type: Superiority or Other; p < 0.001, Log Rank — No adjustments for multiple comparisons were made for this endpoint; Stratified by history of diabetes and country. 2-sided test
Statistical Analysis 2: Comparison: Cinacalcet vs Placebo; Test type: Superiority or Other; Regression, Cox; Stratified by history of diabetes and country; Hazard Ratio (HR) = 0.44, 95% CI 2-sided [0.36 to 0.54] — HR is cinacalcet vs placebo

ADVERSE EVENTS:
Time Frame: Average 24 months
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events. The number of participants at risk includes subjects who received at least 1 dose of investigational product.
Arm/Group | Placebo | Cinacalcet
Serious Adverse Events (participants affected / at risk) | 1351/1923 | 1338/1938
Other Adverse Events (participants affected / at risk) | 1220/1923 | 1444/1938
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=1923) | Cinacalcet (N=1938)
Anaemia (Blood and lymphatic system disorders) | 35 | 42
Coagulopathy (Blood and lymphatic system disorders) | 1 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Haemolysis (Blood and lymphatic system disorders) | 1 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 4 | 5
Haemorrhagic disorder (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 4
Leukopenia (Blood and lymphatic system disorders) | 1 | 2
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 1
Lymphatic disorder (Blood and lymphatic system disorders) | 1 | 0
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 2
Pancytopenia (Blood and lymphatic system disorders) | 4 | 2
Polycythaemia (Blood and lymphatic system disorders) | 1 | 1
Retroperitoneal lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Splenic infarction (Blood and lymphatic system disorders) | 1 | 0
Splenomegaly (Blood and lymphatic system disorders) | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 3
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 14 | 6
Acute left ventricular failure (Cardiac disorders) | 3 | 0
Acute myocardial infarction (Cardiac disorders) | 34 | 47
Angina pectoris (Cardiac disorders) | 42 | 36
Angina unstable (Cardiac disorders) | 42 | 52
Aortic valve incompetence (Cardiac disorders) | 1 | 1
Aortic valve stenosis (Cardiac disorders) | 2 | 7
Arrhythmia (Cardiac disorders) | 17 | 8
Arrhythmia supraventricular (Cardiac disorders) | 2 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 8 | 4
Atrial fibrillation (Cardiac disorders) | 68 | 56
Atrial flutter (Cardiac disorders) | 10 | 12
Atrial tachycardia (Cardiac disorders) | 0 | 1
Atrioventricular block (Cardiac disorders) | 3 | 5
Atrioventricular block complete (Cardiac disorders) | 7 | 6
Atrioventricular block first degree (Cardiac disorders) | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 2 | 1
Atrioventricular dissociation (Cardiac disorders) | 1 | 1
Bradyarrhythmia (Cardiac disorders) | 2 | 2
Bradycardia (Cardiac disorders) | 9 | 12
Bundle branch block (Cardiac disorders) | 0 | 1
Bundle branch block right (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 57 | 60
Cardiac disorder (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 90 | 74
Cardiac failure acute (Cardiac disorders) | 4 | 6
Cardiac failure chronic (Cardiac disorders) | 5 | 4
Cardiac failure congestive (Cardiac disorders) | 86 | 64
Cardiac flutter (Cardiac disorders) | 1 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 1
Cardiac valve disease (Cardiac disorders) | 2 | 0
Cardio-respiratory arrest (Cardiac disorders) | 21 | 27
Cardiogenic shock (Cardiac disorders) | 8 | 12
Cardiomyopathy (Cardiac disorders) | 7 | 6
Cardiopulmonary failure (Cardiac disorders) | 6 | 6
Cardiovascular disorder (Cardiac disorders) | 0 | 1
Cardiovascular insufficiency (Cardiac disorders) | 1 | 1
Congestive cardiomyopathy (Cardiac disorders) | 4 | 1
Coronary artery disease (Cardiac disorders) | 23 | 28
Coronary artery insufficiency (Cardiac disorders) | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 1 | 1
Coronary artery stenosis (Cardiac disorders) | 4 | 5
Diastolic dysfunction (Cardiac disorders) | 1 | 1
Dilatation ventricular (Cardiac disorders) | 0 | 1
Gastrocardiac syndrome (Cardiac disorders) | 1 | 0
Heart valve stenosis (Cardiac disorders) | 1 | 0
Hypertensive heart disease (Cardiac disorders) | 2 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 4 | 2
Left ventricular dysfunction (Cardiac disorders) | 0 | 2
Left ventricular failure (Cardiac disorders) | 6 | 1
Left ventricular hypertrophy (Cardiac disorders) | 1 | 0
Mitral valve calcification (Cardiac disorders) | 0 | 1
Mitral valve disease (Cardiac disorders) | 0 | 2
Mitral valve incompetence (Cardiac disorders) | 3 | 2
Mitral valve stenosis (Cardiac disorders) | 3 | 2
Myocardial infarction (Cardiac disorders) | 105 | 109
Myocardial ischaemia (Cardiac disorders) | 10 | 11
Myocarditis (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 4 | 6
Pericardial effusion (Cardiac disorders) | 5 | 8
Pericardial haemorrhage (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 2 | 3
Pericarditis uraemic (Cardiac disorders) | 2 | 2
Pulseless electrical activity (Cardiac disorders) | 5 | 2
Right ventricular failure (Cardiac disorders) | 1 | 2
Sick sinus syndrome (Cardiac disorders) | 3 | 3
Sinus bradycardia (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 2
Supraventricular extrasystoles (Cardiac disorders) | 0 | 1
Supraventricular tachyarrhythmia (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 6 | 6
Tachyarrhythmia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 6 | 6
Tricuspid valve incompetence (Cardiac disorders) | 1 | 1
Tricuspid valve stenosis (Cardiac disorders) | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 5 | 3
Ventricular extrasystoles (Cardiac disorders) | 1 | 1
Ventricular failure (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 9 | 6
Ventricular tachyarrhythmia (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 5 | 12
Adenomatous polyposis coli (Congenital, familial and genetic disorders) | 0 | 1
Congenital cystic disease of liver (Congenital, familial and genetic disorders) | 1 | 0
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 3 | 6
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 1 | 2
Left ventricle outflow tract obstruction (Congenital, familial and genetic disorders) | 0 | 1
Aural polyp (Ear and labyrinth disorders) | 1 | 0
Deafness unilateral (Ear and labyrinth disorders) | 1 | 0
Meniere's disease (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 2 | 4
Vertigo positional (Ear and labyrinth disorders) | 0 | 1
Vestibular disorder (Ear and labyrinth disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Goitre (Endocrine disorders) | 1 | 0
Hyperparathyroidism (Endocrine disorders) | 86 | 23
Hyperparathyroidism secondary (Endocrine disorders) | 41 | 12
Hyperparathyroidism tertiary (Endocrine disorders) | 8 | 2
Hyperthyroidism (Endocrine disorders) | 2 | 1
Parathyroid disorder (Endocrine disorders) | 1 | 0
Parathyroid gland enlargement (Endocrine disorders) | 1 | 2
Parathyroid haemorrhage (Endocrine disorders) | 1 | 0
Secondary hyperthyroidism (Endocrine disorders) | 1 | 0
Thyroid cyst (Endocrine disorders) | 0 | 1
Thyroiditis (Endocrine disorders) | 0 | 1
Age-related macular degeneration (Eye disorders) | 0 | 1
Cataract (Eye disorders) | 5 | 8
Cataract cortical (Eye disorders) | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 2
Diabetic retinopathy (Eye disorders) | 0 | 1
Diplopia (Eye disorders) | 1 | 1
Exophthalmos (Eye disorders) | 0 | 1
Eye haemorrhage (Eye disorders) | 0 | 3
Glaucoma (Eye disorders) | 1 | 0
Keratitis (Eye disorders) | 1 | 0
Optic atrophy (Eye disorders) | 0 | 1
Optic ischaemic neuropathy (Eye disorders) | 1 | 0
Papilloedema (Eye disorders) | 1 | 0
Photopsia (Eye disorders) | 1 | 0
Retinal artery occlusion (Eye disorders) | 1 | 0
Retinal detachment (Eye disorders) | 0 | 3
Retinal vein thrombosis (Eye disorders) | 0 | 1
Retinopathy hypertensive (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 0
Visual impairment (Eye disorders) | 0 | 1
Vitreous haemorrhage (Eye disorders) | 1 | 2
Abdominal discomfort (Gastrointestinal disorders) | 3 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 4 | 4
Abdominal hernia obstructive (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 42 | 33
Abdominal pain lower (Gastrointestinal disorders) | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 5
Abdominal rigidity (Gastrointestinal disorders) | 0 | 1
Abdominal strangulated hernia (Gastrointestinal disorders) | 0 | 2
Anal fistula (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 7 | 3
Barrett's oesophagus (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 7 | 5
Colitis ischaemic (Gastrointestinal disorders) | 3 | 9
Colitis ulcerative (Gastrointestinal disorders) | 1 | 1
Colonic polyp (Gastrointestinal disorders) | 7 | 2
Colonic pseudo-obstruction (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 8
Dental caries (Gastrointestinal disorders) | 1 | 0
Diabetic gastroparesis (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 24 | 32
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 | 0
Dieulafoy's vascular malformation (Gastrointestinal disorders) | 0 | 1
Diverticular perforation (Gastrointestinal disorders) | 1 | 2
Diverticulum (Gastrointestinal disorders) | 0 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 2 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 0
Duodenal perforation (Gastrointestinal disorders) | 2 | 0
Duodenal ulcer (Gastrointestinal disorders) | 4 | 7
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Duodenitis (Gastrointestinal disorders) | 4 | 2
Duodenitis haemorrhagic (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 3
Dysphagia (Gastrointestinal disorders) | 2 | 3
Enteritis (Gastrointestinal disorders) | 1 | 5
Enterocolitis (Gastrointestinal disorders) | 1 | 1
Erosive duodenitis (Gastrointestinal disorders) | 1 | 1
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 1
Faecaloma (Gastrointestinal disorders) | 1 | 3
Faeces discoloured (Gastrointestinal disorders) | 1 | 1
Gastric antral vascular ectasia (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 4 | 1
Gastric hypermotility (Gastrointestinal disorders) | 0 | 1
Gastric perforation (Gastrointestinal disorders) | 2 | 0
Gastric polyps (Gastrointestinal disorders) | 1 | 1
Gastric ulcer (Gastrointestinal disorders) | 6 | 12
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 2
Gastritis (Gastrointestinal disorders) | 15 | 10
Gastritis erosive (Gastrointestinal disorders) | 6 | 5
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 1
Gastroduodenitis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 0 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 53 | 54
Gastrointestinal hypomotility (Gastrointestinal disorders) | 1 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 | 2
Gastrointestinal necrosis (Gastrointestinal disorders) | 2 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 | 0
Gastrointestinal oedema (Gastrointestinal disorders) | 1 | 0
Gastrointestinal perforation (Gastrointestinal disorders) | 2 | 0
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 4
Haematemesis (Gastrointestinal disorders) | 3 | 5
Haematochezia (Gastrointestinal disorders) | 2 | 2
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2 | 2
Haemorrhoids (Gastrointestinal disorders) | 2 | 5
Hernial eventration (Gastrointestinal disorders) | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 1 | 2
Ileus (Gastrointestinal disorders) | 4 | 6
Impaired gastric emptying (Gastrointestinal disorders) | 2 | 6
Inguinal hernia (Gastrointestinal disorders) | 2 | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Intestinal infarction (Gastrointestinal disorders) | 3 | 3
Intestinal ischaemia (Gastrointestinal disorders) | 6 | 9
Intestinal mass (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 3 | 5
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Intestinal polyp (Gastrointestinal disorders) | 1 | 0
Intestinal strangulation (Gastrointestinal disorders) | 1 | 0
Intestinal ulcer (Gastrointestinal disorders) | 0 | 1
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1
Ischaemic gastritis (Gastrointestinal disorders) | 0 | 1
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Large intestinal ulcer (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 4 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 | 3
Lumbar hernia (Gastrointestinal disorders) | 0 | 1
Mechanical ileus (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 2 | 3
Mesenteric artery stenosis (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 16 | 20
Necrotising colitis (Gastrointestinal disorders) | 0 | 1
Oesophageal achalasia (Gastrointestinal disorders) | 0 | 1
Oesophageal disorder (Gastrointestinal disorders) | 1 | 0
Oesophageal food impaction (Gastrointestinal disorders) | 0 | 1
Oesophageal haemorrhage (Gastrointestinal disorders) | 1 | 0
Oesophageal perforation (Gastrointestinal disorders) | 0 | 1
Oesophageal rupture (Gastrointestinal disorders) | 1 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 2 | 0
Oesophagitis (Gastrointestinal disorders) | 3 | 6
Oesophagitis haemorrhagic (Gastrointestinal disorders) | 0 | 1
Pancreatic mass (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 11 | 10
Pancreatitis acute (Gastrointestinal disorders) | 9 | 7
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 2
Peptic ulcer (Gastrointestinal disorders) | 2 | 1
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Peritoneal disorder (Gastrointestinal disorders) | 1 | 0
Portal hypertensive enteropathy (Gastrointestinal disorders) | 1 | 0
Portal hypertensive gastropathy (Gastrointestinal disorders) | 1 | 0
Proctitis (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 12 | 12
Rectal ulcer (Gastrointestinal disorders) | 1 | 1
Rectal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Retroperitoneal haematoma (Gastrointestinal disorders) | 2 | 2
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 1
Retroperitoneal mass (Gastrointestinal disorders) | 1 | 0
Short-bowel syndrome (Gastrointestinal disorders) | 0 | 1
Sigmoiditis (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 5
Stomach mass (Gastrointestinal disorders) | 0 | 1
Stress ulcer (Gastrointestinal disorders) | 0 | 1
Subileus (Gastrointestinal disorders) | 0 | 1
Tooth loss (Gastrointestinal disorders) | 0 | 1
Tooth socket haemorrhage (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 2 | 0
Umbilical hernia (Gastrointestinal disorders) | 3 | 1
Umbilical hernia, obstructive (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 8 | 11
Uraemic gastropathy (Gastrointestinal disorders) | 1 | 0
Varices oesophageal (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 23 | 33
Adverse drug reaction (General disorders) | 1 | 1
Asthenia (General disorders) | 20 | 15
Calcinosis (General disorders) | 2 | 0
Catheter site haematoma (General disorders) | 1 | 3
Catheter site haemorrhage (General disorders) | 5 | 3
Catheter site pain (General disorders) | 0 | 1
Catheter site swelling (General disorders) | 0 | 1
Chest discomfort (General disorders) | 3 | 4
Chest pain (General disorders) | 53 | 51
Chills (General disorders) | 2 | 4
Condition aggravated (General disorders) | 1 | 0
Cyst (General disorders) | 1 | 1
Death (General disorders) | 38 | 38
Device breakage (General disorders) | 1 | 0
Device dislocation (General disorders) | 1 | 2
Device failure (General disorders) | 2 | 0
Device malfunction (General disorders) | 2 | 2
Device occlusion (General disorders) | 1 | 2
Drug intolerance (General disorders) | 0 | 1
Drug withdrawal syndrome (General disorders) | 0 | 1
Face oedema (General disorders) | 1 | 1
Fat necrosis (General disorders) | 0 | 1
Fatigue (General disorders) | 3 | 1
Feeling abnormal (General disorders) | 1 | 0
Gait disturbance (General disorders) | 2 | 0
General physical health deterioration (General disorders) | 8 | 7
Granuloma (General disorders) | 1 | 0
Hernia (General disorders) | 0 | 1
Hernia obstructive (General disorders) | 4 | 0
Hernia pain (General disorders) | 0 | 1
Hyperthermia (General disorders) | 1 | 2
Hypothermia (General disorders) | 2 | 2
Impaired healing (General disorders) | 10 | 5
Implant site effusion (General disorders) | 1 | 0
Implant site haematoma (General disorders) | 0 | 1
Inflammation (General disorders) | 1 | 0
Influenza like illness (General disorders) | 0 | 1
Infusion site thrombosis (General disorders) | 1 | 0
Ischaemic ulcer (General disorders) | 4 | 0
Localised oedema (General disorders) | 0 | 1
Malaise (General disorders) | 4 | 4
Medical device complication (General disorders) | 17 | 9
Multi-organ failure (General disorders) | 5 | 8
Necrosis (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 23 | 27
Oedema (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 5 | 4
Organ failure (General disorders) | 0 | 1
Pain (General disorders) | 4 | 1
Pelvic mass (General disorders) | 0 | 1
Polyserositis (General disorders) | 1 | 0
Precancerous mucosal lesion (General disorders) | 0 | 1
Pyrexia (General disorders) | 35 | 42
Spinal pain (General disorders) | 1 | 2
Sudden cardiac death (General disorders) | 7 | 7
Sudden death (General disorders) | 26 | 22
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Thrombosis in device (General disorders) | 5 | 4
Ulcer (General disorders) | 2 | 1
Ulcer haemorrhage (General disorders) | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 3
Biliary colic (Hepatobiliary disorders) | 2 | 0
Biliary dyskinesia (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 2 | 3
Cholangitis acute (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 10 | 9
Cholecystitis acute (Hepatobiliary disorders) | 5 | 7
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 12 | 16
Cholestasis (Hepatobiliary disorders) | 1 | 2
Chronic hepatic failure (Hepatobiliary disorders) | 1 | 0
Gallbladder perforation (Hepatobiliary disorders) | 1 | 0
Gallbladder polyp (Hepatobiliary disorders) | 0 | 2
Hepatic cirrhosis (Hepatobiliary disorders) | 3 | 2
Hepatic congestion (Hepatobiliary disorders) | 1 | 0
Hepatic cyst ruptured (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 3 | 2
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Hepatic lesion (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 2 | 0
Hepatitis toxic (Hepatobiliary disorders) | 2 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 1
Liver disorder (Hepatobiliary disorders) | 1 | 0
Amyloidosis (Immune system disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 3 | 1
Contrast media allergy (Immune system disorders) | 1 | 0
Dialysis amyloidosis (Immune system disorders) | 1 | 1
Kidney transplant rejection (Immune system disorders) | 3 | 6
Transplant rejection (Immune system disorders) | 1 | 1
Abdominal abscess (Infections and infestations) | 1 | 2
Abdominal sepsis (Infections and infestations) | 3 | 0
Abdominal wall abscess (Infections and infestations) | 1 | 4
Abdominal wall infection (Infections and infestations) | 1 | 0
Abscess (Infections and infestations) | 2 | 3
Abscess intestinal (Infections and infestations) | 2 | 1
Abscess limb (Infections and infestations) | 5 | 9
Abscess neck (Infections and infestations) | 0 | 1
Abscess of eyelid (Infections and infestations) | 0 | 1
Abscess oral (Infections and infestations) | 0 | 1
Acute sinusitis (Infections and infestations) | 0 | 1
Amoebic dysentery (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 4 | 6
Appendicitis perforated (Infections and infestations) | 0 | 1
Arteriosclerotic gangrene (Infections and infestations) | 0 | 1
Arteriovenous fistula site infection (Infections and infestations) | 15 | 10
Arteriovenous graft site infection (Infections and infestations) | 14 | 25
Arthritis bacterial (Infections and infestations) | 2 | 4
Arthritis infective (Infections and infestations) | 0 | 2
Bacteraemia (Infections and infestations) | 24 | 27
Bacterial infection (Infections and infestations) | 0 | 1
Bacterial sepsis (Infections and infestations) | 2 | 1
Bartholin's abscess (Infections and infestations) | 1 | 0
Biliary sepsis (Infections and infestations) | 1 | 1
Biliary tract infection (Infections and infestations) | 0 | 1
Breast cellulitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 25 | 26
Bronchitis bacterial (Infections and infestations) | 1 | 0
Bronchitis viral (Infections and infestations) | 1 | 1
Bronchopneumonia (Infections and infestations) | 7 | 5
Carbuncle (Infections and infestations) | 2 | 0
Catheter site cellulitis (Infections and infestations) | 0 | 2
Catheter site infection (Infections and infestations) | 6 | 6
Cellulitis (Infections and infestations) | 38 | 29
Cellulitis gangrenous (Infections and infestations) | 1 | 0
Cellulitis orbital (Infections and infestations) | 0 | 1
Cellulitis staphylococcal (Infections and infestations) | 1 | 0
Chest wall abscess (Infections and infestations) | 1 | 0
Clostridial infection (Infections and infestations) | 1 | 3
Clostridium colitis (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 7 | 9
Cystitis (Infections and infestations) | 2 | 2
Dengue fever (Infections and infestations) | 0 | 2
Dermo-hypodermitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 28 | 29
Device related sepsis (Infections and infestations) | 18 | 15
Diabetic foot infection (Infections and infestations) | 5 | 1
Diabetic gangrene (Infections and infestations) | 2 | 1
Disseminated tuberculosis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 8 | 9
Ear infection (Infections and infestations) | 1 | 0
Embolic pneumonia (Infections and infestations) | 1 | 0
Emphysematous cystitis (Infections and infestations) | 1 | 0
Empyema (Infections and infestations) | 3 | 2
Endocarditis (Infections and infestations) | 10 | 13
Endocarditis bacterial (Infections and infestations) | 5 | 2
Endocarditis staphylococcal (Infections and infestations) | 1 | 1
Enteritis infectious (Infections and infestations) | 1 | 2
Enterobacter bacteraemia (Infections and infestations) | 1 | 2
Enterobacter pneumonia (Infections and infestations) | 0 | 1
Enterobacter sepsis (Infections and infestations) | 0 | 3
Enterococcal bacteraemia (Infections and infestations) | 2 | 3
Enterococcal infection (Infections and infestations) | 0 | 1
Enterocolitis bacterial (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 2
Erysipelas (Infections and infestations) | 8 | 8
Escherichia bacteraemia (Infections and infestations) | 0 | 1
Escherichia infection (Infections and infestations) | 1 | 0
Escherichia sepsis (Infections and infestations) | 2 | 2
Extradural abscess (Infections and infestations) | 2 | 1
Eye infection (Infections and infestations) | 0 | 2
Fungaemia (Infections and infestations) | 1 | 1
Fungal oesophagitis (Infections and infestations) | 0 | 1
Furuncle (Infections and infestations) | 2 | 0
Gangrene (Infections and infestations) | 42 | 38
Gas gangrene (Infections and infestations) | 0 | 1
Gastric infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 20 | 24
Gastroenteritis clostridial (Infections and infestations) | 1 | 1
Gastroenteritis norovirus (Infections and infestations) | 1 | 1
Gastroenteritis salmonella (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 4 | 8
Giardiasis (Infections and infestations) | 0 | 1
Graft infection (Infections and infestations) | 6 | 2
Groin abscess (Infections and infestations) | 1 | 0
H1N1 influenza (Infections and infestations) | 1 | 3
Haematoma infection (Infections and infestations) | 0 | 2
Haemophilus infection (Infections and infestations) | 0 | 2
Helicobacter infection (Infections and infestations) | 0 | 1
Hepatitis B (Infections and infestations) | 1 | 1
Hepatitis C (Infections and infestations) | 0 | 2
Herpes zoster (Infections and infestations) | 2 | 4
Herpes zoster ophthalmic (Infections and infestations) | 1 | 0
Implant site infection (Infections and infestations) | 0 | 1
Incision site infection (Infections and infestations) | 1 | 0
Infected fistula (Infections and infestations) | 0 | 3
Infected skin ulcer (Infections and infestations) | 7 | 5
Infection (Infections and infestations) | 11 | 11
Infectious peritonitis (Infections and infestations) | 0 | 1
Infectious pleural effusion (Infections and infestations) | 1 | 0
Infective aneurysm (Infections and infestations) | 0 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 1
Infective tenosynovitis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 2 | 4
Intervertebral discitis (Infections and infestations) | 4 | 4
Joint abscess (Infections and infestations) | 0 | 1
Kidney infection (Infections and infestations) | 1 | 0
Klebsiella bacteraemia (Infections and infestations) | 0 | 1
Laryngitis (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 2 | 2
Lobar pneumonia (Infections and infestations) | 17 | 14
Localised infection (Infections and infestations) | 17 | 11
Lower respiratory tract infection (Infections and infestations) | 8 | 11
Lower respiratory tract infection bacterial (Infections and infestations) | 0 | 1
Lower respiratory tract infection viral (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 4 | 3
Lymph gland infection (Infections and infestations) | 1 | 0
Meningitis (Infections and infestations) | 2 | 1
Meningitis bacterial (Infections and infestations) | 0 | 1
Meningitis cryptococcal (Infections and infestations) | 0 | 1
Meningitis viral (Infections and infestations) | 0 | 1
Morganella infection (Infections and infestations) | 1 | 0
Nasal abscess (Infections and infestations) | 0 | 1
Necrotising fasciitis (Infections and infestations) | 2 | 2
Oesophageal candidiasis (Infections and infestations) | 2 | 1
Orchitis (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 26 | 15
Osteomyelitis chronic (Infections and infestations) | 1 | 0
Otitis externa (Infections and infestations) | 1 | 0
Otitis externa bacterial (Infections and infestations) | 1 | 0
Parotitis (Infections and infestations) | 1 | 0
Perineal abscess (Infections and infestations) | 1 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 1
Perirectal abscess (Infections and infestations) | 0 | 2
Peritoneal abscess (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 7 | 9
Peritonitis bacterial (Infections and infestations) | 3 | 1
Peritonsillar abscess (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 3 | 1
Pilonidal cyst (Infections and infestations) | 0 | 1
Pleural infection (Infections and infestations) | 1 | 0
Pneumococcal bacteraemia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 171 | 118
Pneumonia bacterial (Infections and infestations) | 1 | 1
Pneumonia cytomegaloviral (Infections and infestations) | 1 | 0
Pneumonia escherichia (Infections and infestations) | 0 | 1
Pneumonia fungal (Infections and infestations) | 0 | 1
Pneumonia pneumococcal (Infections and infestations) | 1 | 0
Pneumonia primary atypical (Infections and infestations) | 0 | 2
Pneumonia staphylococcal (Infections and infestations) | 1 | 1
Pneumonia streptococcal (Infections and infestations) | 2 | 0
Pneumonia viral (Infections and infestations) | 0 | 2
Post procedural infection (Infections and infestations) | 0 | 1
Post procedural pneumonia (Infections and infestations) | 0 | 1
Post procedural sepsis (Infections and infestations) | 1 | 0
Postoperative abscess (Infections and infestations) | 1 | 3
Postoperative wound infection (Infections and infestations) | 14 | 7
Pseudomembranous colitis (Infections and infestations) | 2 | 0
Pseudomonas infection (Infections and infestations) | 0 | 1
Pulmonary sepsis (Infections and infestations) | 2 | 1
Pulmonary tuberculosis (Infections and infestations) | 0 | 1
Purulent discharge (Infections and infestations) | 1 | 0
Pyelocystitis (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 3 | 9
Pyelonephritis acute (Infections and infestations) | 0 | 2
Pyelonephritis chronic (Infections and infestations) | 2 | 0
Pyonephrosis (Infections and infestations) | 1 | 1
Rectal abscess (Infections and infestations) | 0 | 1
Renal abscess (Infections and infestations) | 1 | 1
Renal cyst infection (Infections and infestations) | 1 | 2
Respiratory tract infection (Infections and infestations) | 8 | 8
Respiratory tract infection bacterial (Infections and infestations) | 0 | 1
Respiratory tract infection fungal (Infections and infestations) | 1 | 1
Respiratory tract infection viral (Infections and infestations) | 0 | 1
Retroperitoneal abscess (Infections and infestations) | 1 | 1
Scrotal abscess (Infections and infestations) | 0 | 1
Scrotal gangrene (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 111 | 123
Sepsis syndrome (Infections and infestations) | 3 | 2
Septic shock (Infections and infestations) | 35 | 35
Serratia bacteraemia (Infections and infestations) | 0 | 1
Serratia sepsis (Infections and infestations) | 1 | 0
Shunt infection (Infections and infestations) | 3 | 3
Sinusitis (Infections and infestations) | 2 | 2
Skin infection (Infections and infestations) | 3 | 2
Soft tissue infection (Infections and infestations) | 1 | 0
Staphylococcal abscess (Infections and infestations) | 2 | 0
Staphylococcal bacteraemia (Infections and infestations) | 8 | 9
Staphylococcal infection (Infections and infestations) | 9 | 14
Staphylococcal osteomyelitis (Infections and infestations) | 0 | 2
Staphylococcal sepsis (Infections and infestations) | 7 | 12
Streptococcal bacteraemia (Infections and infestations) | 1 | 1
Streptococcal sepsis (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 4 | 6
Systemic candida (Infections and infestations) | 2 | 0
Testicular abscess (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 0 | 1
Tracheobronchitis (Infections and infestations) | 2 | 1
Tuberculosis (Infections and infestations) | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 7
Urethritis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 23 | 18
Urinary tract infection enterococcal (Infections and infestations) | 1 | 0
Urinary tract infection fungal (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 3 | 2
Vestibular neuronitis (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 2 | 5
Viral pharyngitis (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 10 | 7
Wound infection bacterial (Infections and infestations) | 0 | 1
Wound infection staphylococcal (Infections and infestations) | 1 | 2
Zygomycosis (Infections and infestations) | 0 | 1
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 2
Anastomotic stenosis (Injury, poisoning and procedural complications) | 1 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 5 | 9
Arteriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 10 | 3
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 8 | 13
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 44 | 36
Arteriovenous fistula site haematoma (Injury, poisoning and procedural complications) | 2 | 3
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 23 | 17
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 43 | 49
Arteriovenous graft aneurysm (Injury, poisoning and procedural complications) | 0 | 2
Arteriovenous graft site haematoma (Injury, poisoning and procedural complications) | 2 | 0
Arteriovenous graft site haemorrhage (Injury, poisoning and procedural complications) | 7 | 9
Brain contusion (Injury, poisoning and procedural complications) | 1 | 0
Brain herniation (Injury, poisoning and procedural complications) | 0 | 1
Burns second degree (Injury, poisoning and procedural complications) | 1 | 0
Cardiac valve replacement complication (Injury, poisoning and procedural complications) | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Chest injury (Injury, poisoning and procedural complications) | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 2 | 2
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 2 | 3
Compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 2 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 4
Craniocerebral injury (Injury, poisoning and procedural complications) | 3 | 2
Crush injury (Injury, poisoning and procedural complications) | 1 | 0
Cystitis radiation (Injury, poisoning and procedural complications) | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 1 | 0
Extradural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Eye operation complication (Injury, poisoning and procedural complications) | 0 | 1
Face injury (Injury, poisoning and procedural complications) | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 2 | 1
Fall (Injury, poisoning and procedural complications) | 14 | 8
Femoral neck fracture (Injury, poisoning and procedural complications) | 10 | 8
Femur fracture (Injury, poisoning and procedural complications) | 19 | 13
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 4 | 2
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 3
Foreign body (Injury, poisoning and procedural complications) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 2 | 3
Fractured coccyx (Injury, poisoning and procedural complications) | 0 | 1
Fractured ischium (Injury, poisoning and procedural complications) | 3 | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 1
Graft complication (Injury, poisoning and procedural complications) | 0 | 1
Graft haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Graft thrombosis (Injury, poisoning and procedural complications) | 3 | 7
Haemodialysis-induced symptom (Injury, poisoning and procedural complications) | 3 | 4
Hand fracture (Injury, poisoning and procedural complications) | 3 | 2
Head injury (Injury, poisoning and procedural complications) | 4 | 2
Hip fracture (Injury, poisoning and procedural complications) | 10 | 9
Humerus fracture (Injury, poisoning and procedural complications) | 4 | 2
In-stent coronary artery restenosis (Injury, poisoning and procedural complications) | 0 | 2
Incision site complication (Injury, poisoning and procedural complications) | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 4 | 2
Incisional hernia, obstructive (Injury, poisoning and procedural complications) | 1 | 0
Injury (Injury, poisoning and procedural complications) | 2 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 3 | 5
Joint injury (Injury, poisoning and procedural complications) | 3 | 0
Kidney rupture (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 2 | 1
Ligament injury (Injury, poisoning and procedural complications) | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 4 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 4 | 3
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 2 | 1
Muscle rupture (Injury, poisoning and procedural complications) | 2 | 0
Open fracture (Injury, poisoning and procedural complications) | 1 | 1
Open wound (Injury, poisoning and procedural complications) | 2 | 0
Overdose (Injury, poisoning and procedural complications) | 4 | 6
Patella fracture (Injury, poisoning and procedural complications) | 2 | 2
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 3
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 | 0
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 | 0
Perirenal haematoma (Injury, poisoning and procedural complications) | 1 | 1
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 5 | 3
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 4 | 5
Postoperative adhesion (Injury, poisoning and procedural complications) | 0 | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 1
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 0 | 1
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 | 2
Procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Procedural haemorrhage (Injury, poisoning and procedural complications) | 2 | 1
Procedural hypotension (Injury, poisoning and procedural complications) | 2 | 10
Procedural pain (Injury, poisoning and procedural complications) | 2 | 1
Pubis fracture (Injury, poisoning and procedural complications) | 6 | 1
Radius fracture (Injury, poisoning and procedural complications) | 6 | 3
Renal haematoma (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 13 | 6
Road traffic accident (Injury, poisoning and procedural complications) | 2 | 2
Shunt aneurysm (Injury, poisoning and procedural complications) | 0 | 1
Shunt malfunction (Injury, poisoning and procedural complications) | 4 | 3
Shunt occlusion (Injury, poisoning and procedural complications) | 7 | 10
Shunt stenosis (Injury, poisoning and procedural complications) | 4 | 6
Shunt thrombosis (Injury, poisoning and procedural complications) | 7 | 8
Skull fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal column injury (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 5 | 5
Spinal fracture (Injury, poisoning and procedural complications) | 2 | 2
Splenic rupture (Injury, poisoning and procedural complications) | 0 | 1
Sternal fracture (Injury, poisoning and procedural complications) | 1 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 6 | 8
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Suture rupture (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 14 | 5
Thermal burn (Injury, poisoning and procedural complications) | 2 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 6 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 5 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0
Transplant failure (Injury, poisoning and procedural complications) | 1 | 3
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Traumatic lung injury (Injury, poisoning and procedural complications) | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 3 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 3 | 2
Vascular access complication (Injury, poisoning and procedural complications) | 13 | 15
Vascular graft complication (Injury, poisoning and procedural complications) | 11 | 13
Vascular graft occlusion (Injury, poisoning and procedural complications) | 6 | 8
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 27 | 21
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 6 | 8
Vascular pseudoaneurysm ruptured (Injury, poisoning and procedural complications) | 1 | 1
Venous injury (Injury, poisoning and procedural complications) | 1 | 1
Wound (Injury, poisoning and procedural complications) | 4 | 3
Wound decomposition (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 4
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Wound necrosis (Injury, poisoning and procedural complications) | 1 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 7 | 3
Blood calcium decreased (Investigations) | 0 | 1
Blood culture positive (Investigations) | 2 | 1
Blood parathyroid hormone abnormal (Investigations) | 1 | 0
Blood parathyroid hormone increased (Investigations) | 2 | 2
Blood potassium increased (Investigations) | 1 | 4
Blood pressure increased (Investigations) | 1 | 2
C-reactive protein increased (Investigations) | 0 | 2
Cardioactive drug level increased (Investigations) | 0 | 1
Clostridium test positive (Investigations) | 0 | 1
Coagulation time prolonged (Investigations) | 1 | 1
Coagulation time shortened (Investigations) | 1 | 0
Ejection fraction decreased (Investigations) | 1 | 0
Electrocardiogram ST segment abnormal (Investigations) | 0 | 1
Electrocardiogram ST-T segment abnormal (Investigations) | 0 | 1
Electrocardiogram abnormal (Investigations) | 0 | 2
Electrocardiogram change (Investigations) | 0 | 3
Fibrin D dimer increased (Investigations) | 0 | 1
Haematocrit decreased (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 6
Heart rate increased (Investigations) | 1 | 0
Heart rate irregular (Investigations) | 0 | 1
Influenza virus test positive (Investigations) | 0 | 1
International normalised ratio abnormal (Investigations) | 1 | 0
International normalised ratio decreased (Investigations) | 0 | 1
International normalised ratio fluctuation (Investigations) | 0 | 1
International normalised ratio increased (Investigations) | 1 | 2
Liver function test abnormal (Investigations) | 0 | 1
Myocardial strain (Investigations) | 1 | 0
Pulse absent (Investigations) | 1 | 1
Transaminases increased (Investigations) | 1 | 0
Troponin increased (Investigations) | 4 | 1
Weight decreased (Investigations) | 3 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 3
Cachexia (Metabolism and nutrition disorders) | 3 | 4
Calciphylaxis (Metabolism and nutrition disorders) | 13 | 3
Decreased appetite (Metabolism and nutrition disorders) | 0 | 3
Dehydration (Metabolism and nutrition disorders) | 5 | 6
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 3 | 3
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 3 | 4
Dystrophic calcification (Metabolism and nutrition disorders) | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 5 | 6
Fluid overload (Metabolism and nutrition disorders) | 51 | 40
Fluid retention (Metabolism and nutrition disorders) | 8 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 7 | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 74 | 97
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1
Hypervolaemia (Metabolism and nutrition disorders) | 2 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 8 | 16
Hypoglycaemia (Metabolism and nutrition disorders) | 27 | 34
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 2
Shock hypoglycaemic (Metabolism and nutrition disorders) | 0 | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 11
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 9
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 2
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 1
Chondropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 2
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Fracture delayed union (Musculoskeletal and connective tissue disorders) | 1 | 0
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 1 | 0
High turnover osteopathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 6
Joint destruction (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 4 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 2
Kyphosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Ligamentitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Limb deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 6 | 9
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 | 3
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 | 3
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 2 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 15 | 12
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 4
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 13
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 | 0
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Renal osteodystrophy (Musculoskeletal and connective tissue disorders) | 2 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 2
Scleroderma (Musculoskeletal and connective tissue disorders) | 0 | 1
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal disorder (Musculoskeletal and connective tissue disorders) | 2 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Biliary neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder adenocarcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 7
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 5
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Colon cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Intraocular melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lentigo maligna stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant urinary tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm recurrence (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Paraganglion neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 1
Pleural mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 8
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 6
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Renal oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Urinary tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Vaginal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Vocal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Altered state of consciousness (Nervous system disorders) | 2 | 0
Aphasia (Nervous system disorders) | 0 | 1
Ataxia (Nervous system disorders) | 3 | 0
Autonomic neuropathy (Nervous system disorders) | 0 | 2
Balance disorder (Nervous system disorders) | 2 | 3
Basal ganglia haemorrhage (Nervous system disorders) | 0 | 1
Benign intracranial hypertension (Nervous system disorders) | 1 | 0
Brain oedema (Nervous system disorders) | 3 | 1
Brain stem infarction (Nervous system disorders) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 7 | 1
Carpal tunnel syndrome (Nervous system disorders) | 6 | 4
Cerebellar atrophy (Nervous system disorders) | 1 | 0
Cerebral artery stenosis (Nervous system disorders) | 1 | 0
Cerebral atrophy (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 9 | 10
Cerebral hypoperfusion (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 5
Cerebral ischaemia (Nervous system disorders) | 3 | 2
Cerebrovascular accident (Nervous system disorders) | 66 | 60
Cerebrovascular disorder (Nervous system disorders) | 1 | 1
Clonus (Nervous system disorders) | 0 | 1
Cognitive disorder (Nervous system disorders) | 1 | 1
Coma (Nervous system disorders) | 0 | 3
Convulsion (Nervous system disorders) | 21 | 30
Dementia (Nervous system disorders) | 2 | 1
Demyelinating polyneuropathy (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 5 | 9
Dysarthria (Nervous system disorders) | 1 | 1
Dyskinesia (Nervous system disorders) | 0 | 1
Encephalitis (Nervous system disorders) | 0 | 1
Encephalitis post varicella (Nervous system disorders) | 0 | 1
Encephalomalacia (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 8 | 2
Epilepsy (Nervous system disorders) | 0 | 3
Extrapyramidal disorder (Nervous system disorders) | 1 | 2
Guillain-Barre syndrome (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 3 | 7
Haemorrhagic cerebral infarction (Nervous system disorders) | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 5 | 4
Headache (Nervous system disorders) | 3 | 6
Hemianopia (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 1 | 1
Hemiplegia (Nervous system disorders) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 2 | 2
Hydrocephalus (Nervous system disorders) | 2 | 1
Hypertensive encephalopathy (Nervous system disorders) | 3 | 3
Hypertonia (Nervous system disorders) | 2 | 0
Hypoaesthesia (Nervous system disorders) | 2 | 1
Hypogeusia (Nervous system disorders) | 0 | 1
Hypoglycaemic coma (Nervous system disorders) | 2 | 1
Hypoglycaemic encephalopathy (Nervous system disorders) | 0 | 1
Hypotonia (Nervous system disorders) | 0 | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 | 4
Intracranial hypotension (Nervous system disorders) | 1 | 0
Intracranial pressure increased (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 3 | 8
Lacunar infarction (Nervous system disorders) | 2 | 0
Lethargy (Nervous system disorders) | 2 | 1
Loss of consciousness (Nervous system disorders) | 6 | 5
Mental impairment (Nervous system disorders) | 1 | 1
Metabolic encephalopathy (Nervous system disorders) | 6 | 3
Migraine (Nervous system disorders) | 0 | 2
Myelitis transverse (Nervous system disorders) | 0 | 1
Myelopathy (Nervous system disorders) | 1 | 0
Myoclonus (Nervous system disorders) | 3 | 1
Nerve compression (Nervous system disorders) | 0 | 2
Neuralgia (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 2 | 1
Optic neuritis (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 2
Paraplegia (Nervous system disorders) | 1 | 0
Parkinson's disease (Nervous system disorders) | 1 | 0
Parkinsonism (Nervous system disorders) | 1 | 1
Partial seizures (Nervous system disorders) | 0 | 1
Polyneuropathy (Nervous system disorders) | 2 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 1
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 3
Psychomotor hyperactivity (Nervous system disorders) | 2 | 0
Quadriplegia (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 1
Simple partial seizures (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 2
Speech disorder (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 2 | 1
Spinal cord herniation (Nervous system disorders) | 1 | 0
Status epilepticus (Nervous system disorders) | 2 | 3
Stupor (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 2 | 5
Subdural hygroma (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 32 | 32
Tardive dyskinesia (Nervous system disorders) | 1 | 0
Thalamic infarction (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 12 | 15
Tremor (Nervous system disorders) | 0 | 2
Uraemic encephalopathy (Nervous system disorders) | 0 | 2
Uraemic neuropathy (Nervous system disorders) | 0 | 1
VIIth nerve paralysis (Nervous system disorders) | 2 | 0
Vascular dementia (Nervous system disorders) | 1 | 2
Vascular encephalopathy (Nervous system disorders) | 1 | 1
Vertebral artery occlusion (Nervous system disorders) | 1 | 0
Vertebral artery stenosis (Nervous system disorders) | 1 | 0
Vertebrobasilar insufficiency (Nervous system disorders) | 1 | 0
Aggression (Psychiatric disorders) | 1 | 0
Agitation (Psychiatric disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 2 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 1
Borderline personality disorder (Psychiatric disorders) | 1 | 0
Completed suicide (Psychiatric disorders) | 1 | 1
Confusional state (Psychiatric disorders) | 6 | 8
Conversion disorder (Psychiatric disorders) | 0 | 1
Delirium (Psychiatric disorders) | 3 | 3
Depression (Psychiatric disorders) | 6 | 6
Disorientation (Psychiatric disorders) | 1 | 2
Drug abuse (Psychiatric disorders) | 0 | 2
Hallucination (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 1
Major depression (Psychiatric disorders) | 1 | 2
Mental disorder (Psychiatric disorders) | 1 | 0
Mental disorder due to a general medical condition (Psychiatric disorders) | 2 | 0
Mental status changes (Psychiatric disorders) | 24 | 23
Mood swings (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 2
Restlessness (Psychiatric disorders) | 0 | 1
Schizophrenia (Psychiatric disorders) | 0 | 1
Substance abuse (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 2
Suicide attempt (Psychiatric disorders) | 1 | 0
Azotaemia (Renal and urinary disorders) | 9 | 4
Calculus ureteric (Renal and urinary disorders) | 0 | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 2
Cystitis noninfective (Renal and urinary disorders) | 1 | 1
Haematuria (Renal and urinary disorders) | 10 | 3
Nephrolithiasis (Renal and urinary disorders) | 1 | 2
Obstructive uropathy (Renal and urinary disorders) | 1 | 0
Polyuria (Renal and urinary disorders) | 1 | 1
Renal artery stenosis (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 2
Renal cyst (Renal and urinary disorders) | 2 | 2
Renal cyst haemorrhage (Renal and urinary disorders) | 0 | 1
Renal cyst ruptured (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 6 | 4
Renal failure acute (Renal and urinary disorders) | 2 | 1
Renal failure chronic (Renal and urinary disorders) | 30 | 25
Renal haemorrhage (Renal and urinary disorders) | 1 | 4
Renal impairment (Renal and urinary disorders) | 1 | 0
Renal injury (Renal and urinary disorders) | 0 | 1
Renal mass (Renal and urinary disorders) | 2 | 0
Renal tubular necrosis (Renal and urinary disorders) | 0 | 2
Urethral obstruction (Renal and urinary disorders) | 1 | 0
Urethral prolapse (Renal and urinary disorders) | 0 | 1
Urethral stenosis (Renal and urinary disorders) | 1 | 2
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 | 1
Urinary tract pain (Renal and urinary disorders) | 1 | 0
Vesicoureteric reflux (Renal and urinary disorders) | 1 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 1
Breast haematoma (Reproductive system and breast disorders) | 1 | 0
Breast inflammation (Reproductive system and breast disorders) | 0 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0
Cystocele (Reproductive system and breast disorders) | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0
Epididymitis (Reproductive system and breast disorders) | 0 | 1
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 1
Fibrocystic breast disease (Reproductive system and breast disorders) | 0 | 1
Menometrorrhagia (Reproductive system and breast disorders) | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 5 | 1
Ovarian cyst (Reproductive system and breast disorders) | 2 | 1
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 | 0
Pelvic adhesions (Reproductive system and breast disorders) | 0 | 1
Priapism (Reproductive system and breast disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 3 | 3
Scrotal haematocoele (Reproductive system and breast disorders) | 0 | 1
Scrotal pain (Reproductive system and breast disorders) | 0 | 1
Scrotal swelling (Reproductive system and breast disorders) | 0 | 1
Testicular haemorrhage (Reproductive system and breast disorders) | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 1 | 2
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Vaginal laceration (Reproductive system and breast disorders) | 0 | 1
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 23 | 20
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 12 | 10
Alveolitis fibrosing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 7 | 6
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 16 | 20
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 44 | 47
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 | 10
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 7 | 4
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 11 | 8
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Laryngeal cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngeal ulceration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Lupus pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 18 | 32
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 15 | 14
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 8 | 7
Pulmonary necrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 44 | 39
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 5 | 8
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 40 | 31
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Acute generalised exanthematous pustulosis (Skin and subcutaneous tissue disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Angiodermatitis (Skin and subcutaneous tissue disorders) | 1 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 2 | 3
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 3 | 9
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Dry gangrene (Skin and subcutaneous tissue disorders) | 3 | 3
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 1
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 0 | 1
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 1 | 0
Neurodermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 4 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 3 | 3
Skin necrosis (Skin and subcutaneous tissue disorders) | 2 | 4
Skin ulcer (Skin and subcutaneous tissue disorders) | 21 | 20
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0
Activities of daily living impaired (Social circumstances) | 0 | 1
Homicide (Social circumstances) | 1 | 0
Refusal of treatment by patient (Social circumstances) | 1 | 0
Treatment noncompliance (Social circumstances) | 0 | 1
Incisional drainage (Surgical and medical procedures) | 0 | 1
Intraocular lens implant (Surgical and medical procedures) | 1 | 0
Mechanical ventilation (Surgical and medical procedures) | 1 | 0
Therapy cessation (Surgical and medical procedures) | 4 | 5
Accelerated hypertension (Vascular disorders) | 6 | 4
Air embolism (Vascular disorders) | 1 | 0
Aneurysm (Vascular disorders) | 0 | 1
Aneurysm arteriovenous (Vascular disorders) | 3 | 0
Aneurysm ruptured (Vascular disorders) | 1 | 1
Angiopathy (Vascular disorders) | 0 | 1
Aortic aneurysm (Vascular disorders) | 5 | 0
Aortic aneurysm rupture (Vascular disorders) | 1 | 2
Aortic arteriosclerosis (Vascular disorders) | 1 | 1
Aortic dilatation (Vascular disorders) | 1 | 0
Aortic dissection (Vascular disorders) | 2 | 2
Aortic stenosis (Vascular disorders) | 7 | 6
Arterial disorder (Vascular disorders) | 3 | 2
Arterial haemorrhage (Vascular disorders) | 0 | 1
Arterial insufficiency (Vascular disorders) | 0 | 1
Arterial occlusive disease (Vascular disorders) | 2 | 2
Arterial stenosis (Vascular disorders) | 1 | 3
Arterial stenosis limb (Vascular disorders) | 3 | 2
Arterial thrombosis limb (Vascular disorders) | 2 | 2
Arteriosclerosis (Vascular disorders) | 7 | 7
Arteriovenous fistula (Vascular disorders) | 2 | 0
Arteritis (Vascular disorders) | 0 | 5
Bleeding varicose vein (Vascular disorders) | 1 | 0
Blood pressure inadequately controlled (Vascular disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 4 | 2
Deep vein thrombosis (Vascular disorders) | 6 | 10
Diabetic macroangiopathy (Vascular disorders) | 0 | 1
Diabetic vascular disorder (Vascular disorders) | 0 | 3
Embolism (Vascular disorders) | 1 | 1
Embolism arterial (Vascular disorders) | 1 | 0
Exsanguination (Vascular disorders) | 1 | 1
Extremity necrosis (Vascular disorders) | 8 | 6
Femoral arterial stenosis (Vascular disorders) | 2 | 8
Femoral artery occlusion (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 17 | 10
Haemorrhage (Vascular disorders) | 3 | 5
Haemorrhagic infarction (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 44 | 49
Hypertensive crisis (Vascular disorders) | 28 | 29
Hypertensive emergency (Vascular disorders) | 4 | 12
Hypotension (Vascular disorders) | 52 | 54
Hypovolaemic shock (Vascular disorders) | 5 | 2
Iliac artery occlusion (Vascular disorders) | 0 | 1
Iliac artery stenosis (Vascular disorders) | 2 | 4
Iliac artery thrombosis (Vascular disorders) | 1 | 0
Inferior vena caval occlusion (Vascular disorders) | 1 | 0
Intermittent claudication (Vascular disorders) | 2 | 2
Intra-abdominal haematoma (Vascular disorders) | 1 | 2
Ischaemia (Vascular disorders) | 4 | 1
Ischaemic limb pain (Vascular disorders) | 1 | 2
Jugular vein thrombosis (Vascular disorders) | 4 | 0
Leriche syndrome (Vascular disorders) | 1 | 0
Malignant hypertension (Vascular disorders) | 4 | 6
Necrosis ischaemic (Vascular disorders) | 3 | 1
Neurogenic shock (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 3 | 5
Peripheral arterial occlusive disease (Vascular disorders) | 11 | 13
Peripheral artery aneurysm (Vascular disorders) | 0 | 1
Peripheral embolism (Vascular disorders) | 1 | 1
Peripheral ischaemia (Vascular disorders) | 27 | 16
Peripheral vascular disorder (Vascular disorders) | 27 | 30
Phlebitis (Vascular disorders) | 0 | 2
Poor peripheral circulation (Vascular disorders) | 1 | 1
Shock (Vascular disorders) | 3 | 2
Shock haemorrhagic (Vascular disorders) | 2 | 1
Steal syndrome (Vascular disorders) | 4 | 7
Subclavian artery aneurysm (Vascular disorders) | 0 | 1
Subclavian artery stenosis (Vascular disorders) | 0 | 1
Superior vena cava syndrome (Vascular disorders) | 3 | 7
Systolic hypertension (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 2 | 4
Varicose ulceration (Vascular disorders) | 0 | 2
Varicose vein (Vascular disorders) | 1 | 0
Vascular calcification (Vascular disorders) | 0 | 2
Vascular occlusion (Vascular disorders) | 0 | 1
Vascular stenosis (Vascular disorders) | 3 | 3
Vasculitis (Vascular disorders) | 2 | 0
Vena cava thrombosis (Vascular disorders) | 0 | 1
Venous aneurysm (Vascular disorders) | 0 | 1
Venous insufficiency (Vascular disorders) | 1 | 0
Venous occlusion (Vascular disorders) | 3 | 4
Venous stenosis (Vascular disorders) | 4 | 9
Venous thrombosis (Vascular disorders) | 1 | 1
Venous thrombosis limb (Vascular disorders) | 3 | 1
Wegener's granulomatosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=1923) | Cinacalcet (N=1938)
Anaemia (Blood and lymphatic system disorders) | 96 | 109
Abdominal pain (Gastrointestinal disorders) | 154 | 187
Abdominal pain upper (Gastrointestinal disorders) | 121 | 153
Diarrhoea (Gastrointestinal disorders) | 349 | 376
Dyspepsia (Gastrointestinal disorders) | 89 | 140
Nausea (Gastrointestinal disorders) | 288 | 552
Vomiting (Gastrointestinal disorders) | 247 | 482
Chest pain (General disorders) | 119 | 134
Oedema peripheral (General disorders) | 96 | 117
Pyrexia (General disorders) | 161 | 126
Bronchitis (Infections and infestations) | 121 | 138
Nasopharyngitis (Infections and infestations) | 138 | 157
Upper respiratory tract infection (Infections and infestations) | 119 | 144
Urinary tract infection (Infections and infestations) | 94 | 114
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 107 | 124
Decreased appetite (Metabolism and nutrition disorders) | 67 | 112
Hypocalcaemia (Metabolism and nutrition disorders) | 20 | 206
Arthralgia (Musculoskeletal and connective tissue disorders) | 224 | 158
Back pain (Musculoskeletal and connective tissue disorders) | 146 | 159
Muscle spasms (Musculoskeletal and connective tissue disorders) | 174 | 213
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 125 | 109
Pain in extremity (Musculoskeletal and connective tissue disorders) | 193 | 201
Dizziness (Nervous system disorders) | 86 | 135
Headache (Nervous system disorders) | 182 | 219
Cough (Respiratory, thoracic and mediastinal disorders) | 185 | 225
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 188 | 226
Pruritus (Skin and subcutaneous tissue disorders) | 107 | 103
Hypertension (Vascular disorders) | 160 | 176
Hypotension (Vascular disorders) | 154 | 183

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results aftercompletion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.